CLINICAL TRIAL: NCT03604679
Title: A Multicenter, Open-label, Phase I Study of SyB C-0501(Oral Bendamustine) in Patients With Advanced Solid Tumors:
Brief Title: SyB C-0501(Oral Bendamustine) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017003
Record Dates: First submitted 2018-05-30; First posted 2018-07-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SyB C-0501 (Experimental): SyB C-0501 (Oral Bendamustine) will be administered orally once a day (specified dose). The treatment period of 21 days (Cohort 1; 7 days of administration + 14 days of observation or Cohort 2; 14 days of administration + 7 days of observation or Cohort 3; 21 days of administration) constitutes 1 cycle.
  Part 1: dose escalation to determine MTD, RD and dosing schedule Part 2: dose expansion at RD
  Interventions: Drug: SyB C-0501

INTERVENTIONS:
Drug: SyB C-0501 — Specified dose on specified days
  Other Names: bendamustine hydrochloride

SUMMARY:
This study is an open-label, multicenter, phase 1 study of SyB C-0501 by continuous daily oral administration in patients with advanced solid tumors, who have previously received anticancer therapy and consists of two parts. Part 1 is a dose escalation study to evaluate tolerability of SyB C-0501 in the patients, and to find the maximum tolerated dose (MTD), recommended dose (RD) and optimum dosing schedule. Part 2 is being done to evaluate safety and anti-tumor activity of SyB C-0501 preliminarily at RD, and to assess its target cancer exploratory.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or greater at the time of informed consent
* Part 1: Patients with histologically or cytologically confirmed advanced solid tumors refractory to standard therapies or without standard therapies.
* Part 2: patients with advanced solid tumors* refractory to standard therapies or without standard therapies.

  * *metastatic breast cancer, small cell lung cancer and other tumors decided based on the Part 1 results
* ECOG performance status 0-1
* Patients with adequate bone marrow, liver, renal, cardiac and pulmonary function as assessed by the following:

  * Absolute neutrophil count (ANC) ≥ 1500/μL, who has not received supportive care of treatment with GCS within 2 weeks before the entry
  * Platelet count ≥ 100,000/μL and Hemoglobin ≥ 9g/dL in patients received no blood transfusions within 2 weeks before the study entry
  * Serum creatinine ≤ 1.5 x upper limit normal (ULN) or estimated creatinine clearance ≥ 50 mL/min using Cockcroft-Gault equation
  * Serum total bilirubin ≤ 1.5 x ULN in patients not suffering from Gilbert's syndrome
  * ALT and AST ≤ 3.0 x ULN (≤ 5.0 x ULN if liver lesions)
  * 12-lead ECG normal
  * LVEF ≥ 55% by echocardiography
  * SpO2 ≥ 95% or PaO2 ≥ 65mmHg
* Acute toxicity in prior treatment has recovered to baseline or CTCAE Grade 0-1 except the adverse events that, in the judgment of the investigator or sub-investigator, would not provide safety risks in the study.
* Serum/urine pregnancy tests performed before the study entry are negative.
* Male and female patients of childbearing potential should give their consent to use adequate contraceptive measures during the study and 180 days after completing study treatment.
* Provision of written, signed and dated informed consent by the patient or legally acceptable representative after the receipt of adequate information regarding the study
* Ability to understand participation in the study, visiting/treatment plan, sampling/analyses and other study procedures; and willingness to follow them

Exclusion Criteria:

* Active, uncontrollable or symptomatic metastatic tumors in CNS
* Complications of interstitial lung disease, pulmonary fibrosis and emphysema diagnosed by chest-X ray or CT scan
* Medical history of radiation, idiopathic or drug-induced pneumonitis
* Major surgery within 4 weeks before study entry or planning it within 4 weeks
* Treatment with immunotherapy, therapeutic antibody or biologics within 4 weeks or their 5 half-lives before study entry, whichever is longer
* Treatment with cytocidal chemotherapy or hormonal therapy within 14 days
* Radiotherapy within 4 weeks before study entry
* Palliative radiotherapy to control metastatic bone pain within 7 days before study entry
* Malabsorption syndrome or full/partial gastric resection
* Patients intolerable to oral administration in the judgment of the investigator or sub-investigator
* Patients under following medical treatment

  * Anticancer therapy approved for advanced cancers
  * Study treatment in other clinical trials
* Active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV) detected in blood test
* Lactating women
* Medical history of allergy to the agents similar to the investigational drug such as alkylating agents or purine nucleoside derivatives
* Medical history of allergy to Polyoxyl 40 hydrogenated castor oil or gelatin capsule
* Severe acute or chronic physical/mental condition or laboratory abnormalities which could interfere with evaluation of study treatment or results, or which is likely to progress/worsen due to the participation in the study or administration of SyB C-0501
* Any condition that, in the opinion of the investigator or sub-investigator, makes the patient inappropriate for the study participation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Identification of Dose-Limiting Toxicity (DLT) and Number of Subjects with DLT in Each Cohort/Level | Cycle 1 (Approximately 3 weeks)
  Based on the number of patients with DLT and administration dose in each cohort, recommended dosage will be defined for the following clinical phase. A DLT is defined as an adverse event that occurred during the Cycle 1, for which a causality with the investigational products (IP) cannot be ruled out and meets the DLT criteria of this study.
Adverse Events (Types, Incidence, severity, Relationship to SyB C-0501) | Approximately 2 years

SECONDARY OUTCOMES:
Adverse Events (Types, Incidence, Severity, Relationship to SyB C-0501) | Approximately 4 years
Change of laboratory test values and clinical laboratory abnormal values (Incidence, Severity) | Approximately 4 years
Maximum concentration (Cmax) of unchanged bendamustine in plasma | Day 1, and Day 8 or Day 15 of Cycle 1 (each cycle is 21 days)
Time to maximum concentration (tmax) of unchanged bendamustine in plasma | Day 1, and Day 8 or Day15 of Cycle 1 (each cycle is 21 days)
Area under the concentration-time curve up to the last time point with detectable plasma concentration (AUC0-last) of unchanged bendamustine in plasma | Day 1, and Day 8 or Day 15 of Cycle 1 (each cycle is 21 days)
Area under the concentration-time curve up to infinity (AUC0-inf) of unchanged bendamustine in plasma | Day 1, and Day 8 or Day 15 of Cycle 1 (each cycle is 21 days)
Elimination half-life (t1/2) of unchanged bendamustine in plasma | Day 1, and Day 8 or Day 15 of Cycle 1 (each cycle is 21 days)
Oral clearance (CL/F) of unchanged bendamustine in plasma | Day 1, and Day 8 or Day 15 of Cycle 1 (each cycle is 21 days)
Apparent volume of distribution (Vd/F) of unchanged bendamustine in plasma | Day 1, and Day 8 or Day 15 of Cycle 1 (each cycle is 21 days)
Objective Response Rate (ORR), Clinical benefit rate (CBR) and Progression-Free Survival (PFS) | Approximately 4 years
Change of laboratory test values and clinical laboratory abnormal values (Incidence, Severity) | Approximately 2 years
Objective Response Rate (ORR), Clinical benefit rate (CBR) and Progression-Free Survival (PFS) | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Goto, Study Director — SymBio Pharmaceuticals
Locations (2):
- Japan (2):
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Sayama

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shimizu T, Nakagawa K, Hayashi H, Iwasa T, Kawakami H, Watanabe S, Yamamoto N, Yonemori K, Koyama T, Sato J, Tamura K, Kikuchi K, Akaike K, Takeda S, Takeda M. Oral formulation of bendamustine hydrochloride for patients with advanced solid tumors; a phase 1 study. Invest New Drugs. 2023 Feb;41(1):1-12. doi: 10.1007/s10637-022-01307-6. Epub 2022 Nov 4. PMID 36331674